CLINICAL TRIAL: NCT00784602
Title: Observing Pelvic Organ Prolapse Symptoms And Treatment Outcomes
Status: Terminated | Type: Observational
Why Stopped: Shift in department's research interests
Sponsor: Melissa Fischer, MD (Other)
Collaborators: Corewell Health East (Other)
Responsible Party: Sponsor-Investigator, Melissa Fischer, MD, Principal Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Other Study IDs: 2008-242
Record Dates: First submitted 2008-11-03; First posted 2008-11-04 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Genital Prolapse
Keywords: prolapse; pelvic organ prolapse
MeSH Terms: conditions — Prolapse; Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
To prospectively observe the outcomes of surgical prolapse treatment in terms of urinary, bowel, and sexual function, quality of life, patient satisfaction, cost, and achieving patient determined treatment goals.

DETAILED DESCRIPTION:
Patients meeting the inclusion/exclusion criteria will be identified by reviewing the hospital's surgical boarding list and contacted by phone to obtain informed consent. Once informed consent is obtained, chart review will be conducted here at William Beaumont Hospital and at the physician's office to collect patient information related to their prolapse condition. Prior to surgery, questionnaires will be mailed and completed by the participant and then again at 6 and 12 months after surgery, and then yearly. Questionnaires will assess urinary, bowel, and sexual function, and patient treatment goals, treatment satisfaction, and general health and wellbeing. Completion of the questionnaires will be voluntary, and participants will be followed in this manner until voluntary withdrawal, exclusionary criteria emerge, or death.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Pelvic Organ Prolapse
* Able to provide informed consent
* Able to complete study assessments, per clinician judgment

Exclusion Criteria:

* Age < 21 years
* Currently pregnant or < 6 months post-partum

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with genital prolapse.
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2008-10-29 (Actual); Primary Completion 2016-08-29 (Actual); Study Completion 2016-08-29 (Actual)

PRIMARY OUTCOMES:
Changes in urinary, bowel, and sexual function as measured on the PFDI, PFIQ, and PISQ validated questionnaires | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Fischer, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No